CLINICAL TRIAL: NCT07249801
Title: State-dependent Entrainment of Intrinsic Brain Rhythms to Improve Interregional Functional Coupling.
Brief Title: Closed-loop rTMS-EEG During Visuomotor Integration.
Acronym: SYNC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Kirstin-Friederike Heise, Assistant Professor-Faculty, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00144782; 1P50HD118628-01 (NIH)
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Visuomotor Skills; Brain Lesion (General)
Keywords: visuomotor processing; electroencephalography (EEG); transcranial magnetic stimulation (TMS); eye-hand control
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- state-dependent repetitive transcranial magnetic stimulation (rTMS) (Experimental): Repetitive TMS will be applied to cortical targets based on task-based (visuomotor) brain activation.
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation (rTMS) — rTMS will be applied time-locked to the intrinsic brain rhythms to individually-defined brain regions
  Other Names: non-invasive brain stimulation

SUMMARY:
This pilot study aims at establishing personalized state-based rTMS for precision neurorehabilitation, we designed a within-subject cross-over study to test closed-loop repetitive transcranial magnetic stimulation and electroencephalography (rTMS-EEG) comparing the targeting of two key nodes in the frontoparietal network during bimanual visuomotor force tracking in persons with upper extremity sensorimotor impairment affecting eye-hand control.

DETAILED DESCRIPTION:
There is a need for oscillatory or repetitive neuromodulatory tools and methods that are effective in entraining intrinsic neural rhythms to improve inefficient functional coupling within neural circuits. The goal of the proposed study is to develop a closed-loop application of repetitive transcranial magnetic stimulation (rTMS) and electroencephalography (EEG) suitable for use in multidomain precision neural-circuit based rehabilitation studies that permits the time-locked application of rTMS pulses to the phase of the intrinsic neural oscillation (personalized state-based application) in a defined behavioral context (e.g., goal-directed eye-hand control).

ELIGIBILITY:
Inclusion Criteria:

* adult volunteers (age ≥18 years)
* right-hand dominance (defined with the Edinburg Handedness Scale)
* voluntary whole-hand grip force (Medical Research Council scale for muscle force ≥2)
* capable of repeated grasp and release with 5% of maximum voluntary contraction (standardized with an in-house computer-based assessment involving whole-hand grip force tracking upon visual cues with a digital dynamometer).

Exclusion Criteria:

* presence of any MRI risk factors (such as an electrically, magnetically, mechanically activated metal or nonmetal implant including cardiac pacemaker, intracerebral vascular clips, any other electrically sensitive support system, or claustrophobia)
* presence of any contraindications to repetitive transcranial magnetic stimulation, rTMS (e.g., history of seizures or epileptic activity, currently taking medications that lower seizure thresholds)
* any neurological or psychiatric disorders affecting cognitive function (e.g., established dementia) affecting the ability to understand the purpose of the study and give informed consent or ability to complete cognitive testing
* substance use disorder
* visual impairment that precludes completion of scanner tasks
* uncontrolled hypertension despite treatment
* intake of tricyclic anti-depressants
* musculoskeletal disorders affecting bimanual grasp- and release
* pregnancy (or suspected/possible pregnancy or plan to become pregnant in the short term). If the participant is a woman of childbearing potential, a urine pregnancy test will be performed on a standard basis.
* severe aphasia affecting particularly of receptive nature (NIH Stroke Scale, NIHSS Language subsection ≥2) affecting the ability to understand the purpose of the study and give informed consent
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Change of whole hand grip force precision | 90 minutes
  Force time series will be used to extract two measures for each trial to describe distinct features of visuomotor force adjustment: 1) Root Mean Square Error (RMSE) to characterize the deviation of the actual force from the target force, i.e., over- and undershoot and 2) sample entropy (SmpEn) to quantify the randomness or uncertainty of the sampled force time series. From these measures, the trial-based relative changes in RMSE and SmpEn from baseline (before intervention) will be computed.
Change of functional brain connectivity. | 90 minutes
  Trial-specific phase-based connectivity will be extracted from the electroencephalography (EEG) time series and computed relative to baseline (before intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Kirstin-Friederike Heise, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
We intend to comply with NIH Data Management and Sharing Policy. At this stage, the plan is to share de-identified data and supporting documentation in a manner that protects participant privacy and aligns with institutional guidelines. Specific details regarding the scope of data, timing, and access procedures will be finalized as the study progresses.
Supporting Information: Study Protocol, ICF
Time Frame: After primary analyses, anticipated within 12-24 months after study completion.
Access Criteria: Data will be shared through a secure repository. Requests may require a data use agreement and compliance with institutional and regulatory requirements.